CLINICAL TRIAL: NCT01163110
Title: Phase II Dose of Escalation Design to Investigate the Therapeutic Role of RNA Fragments in the Protection of Platelet Production During Chemotherapy
Brief Title: Study to Investigate the Therapeutic Role of RNA Fragments in Platelet Production During Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Midwestern Regional Medical Center (Other)
Responsible Party: Principal Investigator, James Grutsch, PhD, Midwestern Regional Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTCA04-04
Record Dates: First submitted 2010-07-13; First posted 2010-07-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Thrombocytopenia; Neoplasm; Cancer
MeSH Terms: conditions — Thrombocytopenia; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Realbuild — Patient with chemotherapy induced thrombocytopenia takes RNA fragments orally to accelerate time to platelet recovery

SUMMARY:
The purpose of this study is to measure the therapeutic potential of Escherichia coli (E. coli) and yeast ribosomal Ribonucleic acid (RNA) fragments to maintain the production of platelets in patients undergoing cytotoxic therapy for cancer.

DETAILED DESCRIPTION:
Myelosuppressive chemotherapy has the potential to produce life threatening neutropenia, anemia, and thrombocytopenia. All of these conditions compromise therapeutic dosing which impacts survival as well as quality of life. The introduction of recombinant growth factors has enabled oncologists to minimize or prevent the development of treatment-induced anemia and neutropenia, but the management of chemotherapy-induced thrombocytopenia (CIT) remains a major challenge. American Society of Clinical Oncology (ASCO) guidelines recommend dose reduction in chemotherapy following onset of thrombocytopenia despite data showing full dose, on time, chemotherapy leads to reduced tumor burden and better overall survival [1-3]. Patients with CIT experience potentially life threatening complications, delay in treatment, poorer outcomes, and consume inordinate amounts of health care resources for supportive care [4]. Development of an agent that ameliorates CIT would represent a major breakthrough in cancer treatment.

Platelets are anuclear cell particles that are released into the bloodstream by megakaryocytes located in the bone marrow. The differentiation of megakaryocytes is regulated by an intricate interaction of specific cytokines and growth factors [5]. Bone marrow stromal elements are also critical to the differentiation and release of platelets. Cancer chemotherapy often depletes the stem and progenitor cells involved in platelet proliferation, which leads to a diminution of platelets and temporary interruption of platelet production lasting until stromal elements and megakaryocytes regenerate.

There are several experimental agents targeted to prevent thrombocytopenia. These investigational agents are cytokines involved in the differentiation and production of platelets [6]. Currently, the only agent commercially available for prevention of thrombocytopenia is Neumega, a derivative of IL-11. Data on Neumega (Oprelekin) indicates a shorter duration of chemotherapy-induced thrombocytopenia, but the toxicity profile has prevented its widespread introduction into the clinical setting. Overall, the absence of agents that minimize or reverse CIT continues to severely limit many patients' ability to complete the full schedule of chemotherapy at the doses originally prescribed by treating oncologists [1].

This study is a dose escalation trial investigating the anti-thrombocytopenic benefits and safety of single stranded RNA fragments. The short chain RNA fragments are obtained by controlled degradation of prokaryotic RNA with ribonuclease. Beljanski showed that these RNA fragments act as primers for DNA synthesis in vitro and found that variations in the method of degradation yielded different preparations that prime deoxyribonucleic acid (DNA) synthesis with distinct tissue specificity. The RNA fragments used in this study, when administered orally, localize in the bone marrow where they appear to prime DNA replication in stem cells resulting in proliferation of white blood cells and platelets. Beljanski et al. reported that these specific RNA fragments were effective in restoring normal levels of circulating platelets following drug induced thrombocytopenia [7;8]. Demonstrating the utility of these specific RNA fragments for prevention and treatment of thrombocytopenia among cancer patients undergoing chemotherapy is especially attractive given the absence of the side effects associated with growth factors and hormones.

This trial investigated the efficacy of two RNA preparations-extracted, purified and fragmented according Beljanski's procedure-to ameliorate CIT: one derived from E. coli and the second from yeast (a eukaryote). RNA molecules are present in any diet and can be considered conditional essential nutrients under conditions of physiological stress [9]. Purified RNA prepared by various methods can be found in nutritional products for hospitalized patients and infant formula [9-11]. This clinical trial evaluated the biologic effects of various doses of these specially prepared 'primer' RNA fragments on platelet numbers in cancer patients who have already developed thrombocytopenia while undergoing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 80
* currently receiving chemotherapy with a platelet nadir of less than or equal to 80,000
* Eastern Oncology Oncology Group (ECOG) performance status of 0, 1, 2, 3, and 4
* signed informed consent
* willing to take RealBuild and magnesium supplement and undergoing chemotherapy known to induce thrombocytopenia
* willing to stop benzodiazepines
* must be at least 6 hours post therapeutic heparin dose

Exclusion Criteria:

* life expectancy less than three months
* pregnant women or women of childbearing potential who refuse to use prophylaxis against pregnancy while receiving chemotherapy regimens
* patients know hypersensitive to RNA or its metabolic products
* patients requiring therapeutic heparin or benzodiazepines

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Determine whether E. coli or yeast ribosomal ribonucleic acid (rRNA) fragments prophylactically prevent the development of thrombocytopenia during chemotherapy. | Time to Platelet recovery after nadir

SECONDARY OUTCOMES:
Determine whether E. coli or yeast rRNA fragments accelerate the recovery of platelets in patients undergoing chemotherapy. | Time to platelet transfusion 3 weeks after nadir

CONTACTS AND LOCATIONS:
Overall Officials: Robert Levin, MD, Principal Investigator — Midwestern Regional Medical Center
Locations (1):
- Midwestern Regional Medical Center, Zion, Illinois, United States

REFERENCES:
- [Derived] Levin RD, Daehler M, Grutsch JF, Hall JL, Gupta D, Lis CG. Dose escalation study of an anti-thrombocytopenic agent in patients with chemotherapy induced thrombocytopenia. BMC Cancer. 2010 Oct 19;10:565. doi: 10.1186/1471-2407-10-565. PMID 20955619